CLINICAL TRIAL: NCT02993497
Title: Respiratory Measurement Using Infrared Camera and Respiratory Volume Monitor (ExSpiron 1Xi) for Sedation in Patients Undergoing TURP/TURB Under Spinal Anesthesia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 1-2016-0063
Record Dates: First submitted 2016-12-08; First posted 2016-12-15 (Estimated); Last update posted 2017-11-14 (Actual); Status verified 2017-11

CONDITIONS: Prostate Cancer; Bladder Cancer
MeSH Terms: conditions — Prostatic Neoplasms; Urinary Bladder Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Respiratory monitoring group (Experimental)
  Interventions: Device: Infrared camera; Device: RVM(Respiratory Volume Monitor)

INTERVENTIONS:
Device: Infrared camera — In patients undergoing spinal anesthesia, the respiratory parameters are measured using an Infrared camera.
Device: RVM(Respiratory Volume Monitor) — In patients undergoing spinal anesthesia, the respiratory parameters are measured using an RVM(Respiratory Volume Monitor).
  Other Names: ExSpiron™ 1Xi

SUMMARY:
In patients undergoing spinal anesthesia, the investigators used an Infra-red camera and a respiratory volume monitor to determine the accuracy of the ventilation rate of the infra red camera by measuring the respiratory rate, ventilation volume, and ventilation volume with respiratory volume monitor.

ELIGIBILITY:
Inclusion Criteria:

* An adult male who underwent endoscopic prostatectomy resection with regular surgery
* An adult male who underwent endoscopic bladder resection with regular surgery

Exclusion Criteria:

* Presenting alteration in respiratory function detected by functional analysis of lung volume and capacity- pneumonectomy patient, severe ipsilateral destroyed lung patient
* Inability to understand or perform the procedure
* ASA(American Society of Anesthesiologists) class 4,5

Min Age: 19 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2017-02-05 (Actual); Primary Completion 2017-07-04 (Actual); Study Completion 2017-07-04 (Actual)

PRIMARY OUTCOMES:
The accuracy of breathing measurements | Intraoperative period about 1 hour
  The accuracy of breathing measurements between infrared camera and RVM in patients with spinal anesthesia

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Anesthesiology and Pain Medicine, Anesthesia and Pain Research Institute, Yonsei University College of Medicine, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided